CLINICAL TRIAL: NCT04910178
Title: Evaluating the Effect of Pentoxifylline, Ursodiol, and Empagliflozin on Fatty Liver of Patients With Type-2 Diabetes
Brief Title: Follow-up of NAFLD Patients With MRI-PDFF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Asmaa Abdelfattah Elsayed (Other)
Responsible Party: Sponsor-Investigator, Asmaa Abdelfattah Elsayed, PHD candidate in clinical pharmacy department and PI, Beni-Suef University
Organization: Beni-Suef University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BeniSuef
Record Dates: First submitted 2021-05-25; First posted 2021-06-02 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Diabetes Type 2; NAFLD
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Non-alcoholic Fatty Liver Disease | interventions — empagliflozin; Ursodeoxycholic Acid; Pentoxifylline

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Empa group (Experimental): patients will be given Empagliflozin 25 mg once daily
  Interventions: Drug: Empagliflozin 25 MG
- PTX group (Experimental): patients will be given PTX 400 mg twice daily or 3 times daily
  Interventions: Drug: Pentoxifylline 400 MG
- UDCA group (Experimental): patients will be given UDCA 500 mg twice daily
  Interventions: Drug: Ursodeoxycholic acid
- Placebo (Placebo Comparator): patients will be given a placebo
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Empagliflozin 25 MG — tablets to be taken orally once a day
  Other Names: Jardiance 25mg tablets
  Arms: Empa group
Drug: Ursodeoxycholic acid — tablets to be taken orally twice a day
  Other Names: Ursofalk tablets
  Arms: UDCA group
Drug: Pentoxifylline 400 MG — tablets to be taken orally twice a day
  Other Names: Trental tablets
  Arms: PTX group
Other: placebo — just starch tablets without any active agents
  Arms: Placebo

SUMMARY:
The liver is a key organ in metabolism and contributes to T2DM development and insulin resistance via unclear mechanisms that may involve liver fat accumulation, inflammatory signals, and immune cells are proposed to play an important role in the pathogenesis of both NAFLD and T2DM.

DETAILED DESCRIPTION:
This study aims to define

* The effects of PTX, Empagliflozin as an example of SGLT-2 inhibitors and UDCA on liver biomarkers and liver steatosis in type 2 diabetic patients.
* Studying PTX, Empagliflozin as an example of SGLT-2 inhibitors and UDCA efficacy and safety as add-on therapy in type 2 diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are willing to participate in this study
* Adults aged ≥ 18 years old presented at the clinic with a confirmed diagnosis of T2DM who are on sulfonylurea for the last 6 months at least and diagnosed with NAFLD.

Exclusion Criteria:

* • Patients who refused to participate in this trial

  * Patients diagnosed with Type 1 diabetes
  * Previous history of alcohol intake
  * history of recurrent attacks of ketoacidosis in a diabetic patient
  * Type 2 diabetic patient with kidney dysfunction (estimated eGFR below 60ml/min/1.73m2 or CrCl below 60ml/min) or on dialysis
  * Previous history of taking medication that may alter either drug efficacy (eg, corticosteroids, oral contraceptives, and thiazide diuretics)
  * Evidence of another liver disease (viral hepatitis, drug-induced liver disease, autoimmune hepatitis)
  * Lactating/pregnant female or children ≤ 18
  * Any contraindication for Empagliflozin including:

    1. History of recurrent attacks of UTI or Genital infection in females
    2. History of recurrent foot injuries or infections
    3. Type 2 diabetic patient with CV disease especially NYHA classes III/ IV
    4. Immunocompromised patients or with a history of inflammatory, immunological, or malignant diseases.
  * Any contraindication for PTX including:

    1. Hypersensitivity to PTX
    2. Patients with peptic ulcer disease or tendency for bleeding
  * Any contraindication for UDCA including:

    1. Hypersensitivity to UDCA
    2. Patients with biliary disease or hepatobiliary disease (ascites, jaundice)
    3. Patients with hepatic encephalopathy or gallstone pancreatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Adults aged ≥ 18 years old presented at the clinic with a confirmed diagnosis of T2DM
Enrollment: 80 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
liver fat content (percent) | 6-months
  measured by MRI-PDFF
fatty liver staging (0, I, II, and III) | 6-months
  using ultrasound

SECONDARY OUTCOMES:
Changes in Serum Gamma glutamyl transferase (γ-GT) | 6-months
  IU/l
HbA1c (%) | 6-months
Fasting and 2-hr post-prandial serum glucose (mg/dl) | 6-months
Lipid profile | 6-months
  (serum triglycerides, total cholesterol, LDL, HDL) (mg/dl)
Changes in liver enzymes | 6-months
  AST (IU/l) and ALT (IU/l)
Changes in direct and total bilirubin | 6-months
  (mg/dl)
Changes in total protein and albumin | 6-months
  (g/l)

CONTACTS AND LOCATIONS:
Overall Officials: Asmaa A Elsayed, PhD, Principal Investigator — BUC
Locations (1):
- Minya University Hospital, Minya, Egypt

IPD SHARING:
Plan to Share IPD: No